CLINICAL TRIAL: NCT06557564
Title: Development of a Machine Learning Tool for Non-invasive Diagnosis of Liver Graft Pathology Using TruGraf
Brief Title: Diagnosis of Graft Pathology by TruGraf
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Transplant Genomics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 24-5056
Record Dates: First submitted 2024-08-13; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-06

CONDITIONS: Acute Graft Rejection
Keywords: Liver transplant patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Biospecimen Retention: Samples With DNA — TruGraf measures the difference in gene expression for a precise panel of specific genes that have been empirically determined to discriminate between allografts that are truly healthy (Non-ACR), and those in transplant patients that have acute rejection on biopsy (AR).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Liver Transplant patient will be undergoing liver graft biopsy.: Liver transplant patients will be undergoing liver graft biopsy (for any reason), or have had a liver biopsy within 48 hours of consent.
  Interventions: Genetic: TruGraf liver gene expression

INTERVENTIONS:
Genetic: TruGraf liver gene expression — Blood from the patients undergoing graft liver biopsy will be collected on the day of the liver biopsy, preferable prior to tissue collection or within 48 hours following the biopsy. Two specialized PaxGene tubes containing 2.5mL of blood each will be filled and will be sent to TGI laboratory in USA for processing, storage, and analysis using TGI's proprietary bioinformatics TruGraf will provide UHN with a Liver binary result: ACR or non-ACR. The results data will be batched and sent to UHN at agreed upon timepoints.

SUMMARY:
The goal of this observational study is to to identify different causes of liver diseases or damage in liver transplant patients and develop a machine learning algorithm as a non-invasive tool leveraging gene expression and patient clinical information to classify transplant liver diseases We will collect blood samples of the participants who had undergone or will undergo the liver biopsy as part of standard of care, and use this blood in TruGarf. TruGraf is a non-invasive test that measures differentially expressed genes in the blood of transplant recipients to rule out liver damage. Researcher will collect the biopsy result from the medical record and this will be compared with the TruGarf results.

DETAILED DESCRIPTION:
Given the significant investment of healthcare resources into transplantation, it is critical to identify recipients with graft pathologies such as Acute Cellular Rejection (ACR), NASH, cholestasis, etc. at an earlier stage to implement the appropriate intervention, rather than initiating empiric treatment that could be unsafe. This project will develop a practical Machine learning-based tool based on the results of the TruGraf assay alongside clinical and laboratory data for non-invasive diagnosis of graft pathology. TruGraf is a non-invasive test that measures differentially expressed genes in the blood of transplant recipients to identify patients who are likely to be adequately immunosuppressed and, in doing so, rule out graft damage. TruGraf measures the difference in gene expression for a precise panel of specific genes that have been empirically determined to discriminate between allografts that are truly healthy (Non-ACR), and those in transplant patients that have acute rejection on biopsy (AR). Nevertheless, the exact etiology of graft damage may be difficult to discern for the transplant clinician. The clinical characteristics and history of the liver transplant recipient as well as liver enzyme patterns can provide a pre-test probability of one diagnosis being more likely than the other (Acute cellular rejection, NASH, biliary or viral disease). The proposed tool will leverage our expertise in Machine Learning tools applied to clinical and molecular data (TruGraf assay results) to enable effective clinical implementation of the TruGraf assay.

ELIGIBILITY:
Inclusion Criteria:

1. . Single-organ Liver transplant recipients
2. Male or female, age > 18 years at the time of signing informed consent.
3. Willing and able to provide informed consent.
4. Patients will be undergoing liver graft biopsy (for any reason), or have had a liver biopsy within 48 hours of consent.

Exclusion Criteria:

1. Repeat transplant
2. Recipient of multi organ transplantation
3. Any treatment for graft rejection such as IV steroids has been given before biopsy.
4. Targeted biopsies for diagnosis of malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Liver transplant patient with graft pathology
Sampling Method: Probability Sample
Enrollment: 471 (Estimated)
Dates: Start 2024-07-20 (Actual); Primary Completion 2027-07-20 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Develop and validate a ML-based algorithm | 36 months
  Develop and validate a ML-based algorithm that identifies major graft pathologies using liver biopsy as the reference method.

SECONDARY OUTCOMES:
Identify specific etiologies of ongoing graft damage | 36 months
  Identify specific etiologies of ongoing graft damage by examining TruGraf gene expression array.

CONTACTS AND LOCATIONS:
Overall Officials: Mamatha Bhat, MD, Principal Investigator — UHN
Locations (1):
- Toronto General Hospital -UHN, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data will be collected from EPIC by UHN study team. Patient information will be de-identified, and each participant will be identified by a unique study number. The study investigators and UHN Ethics Board may access all PHI being collected for this study for audit/inspection purposes.
Supporting Information: SAP
Time Frame: 36 months
Access Criteria: At the time of publication, data generated and analyzed as part of this study, including de-identified datasets and gene expression, will be made available in appropriate community-endorsed, public repositories and/or databases. In particular, gene expression data, and the corresponding sex, age, and disease type of each sample will be made available in open-access or controlled-access platforms. This access is subject to restrictions that may be imposed via existing collaboration agreements. No identifiers will leave UHN.